CLINICAL TRIAL: NCT05083039
Title: Observational Program to Study the Preventive Efficacy of the BiVac Polio (Oral Polio Vaccine, Divalent, Live Attenuated of Types 1 and 3 ) Vaccine Against the Incidence of Acute Respiratory Infections, Including COVID-19, Produced by FSBSI "Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products", on Volunteers Aged 18-65
Brief Title: Observational Program, Study the Preventive Efficacy of the BiVac Polio Vaccine Against the Incidence of Acute Respiratory Infections, Including COVID-19
Status: Completed | Type: Observational
Sponsor: Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products (Other Government)
Responsible Party: Sponsor
Other Study IDs: BV-PM-05/20
Record Dates: First submitted 2021-10-18; First posted 2021-10-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Coronavirus Infections; Vaccine; Polio
Keywords: Covid-19; SARS-Cov-2; Coronavirus Infections; Immunobiological medicine
MeSH Terms: conditions — Coronavirus Infections; Poliomyelitis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 750 volunteers who will be vaccinated with the BiVac polio vaccine: Group 1 - 750 volunteers, Vaccine 0.2 ml, post-vaccination observation period of 12 months.
- 750 volunteers who will be given a Placebo.: Group 2 - 750 volunteers, Vaccine 0.2ml, post-vaccination observation period of 12 months.

SUMMARY:
Observational program, double-blind, placebo-controlled to study the preventive efficacy of the BiVac polio (Oral polio vaccine, divalent, live attenuated of types 1 and 3 vaccine against the incidence of acute respiratory infections, including COVID-19

DETAILED DESCRIPTION:
To carry out a comparative assessment of the indices of humoral, cellular immunity and cytokine profile in patients with acute respiratory infections.

Current Program Population: 1500 healthy male and female volunteers, aged of between 18 and 65 will be included in the program.

All included volunteers will be divided into groups:

Group 1 - 750 volunteers who will be vaccinated with BiVac polio vaccine; post-vaccination observation period of 12 months.

Group 2 - 750 volunteers, placebo will be administered, post-vaccination observation period of 12 months.

The probability of getting into one of the two groups for each volunteer will be 50%.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must meet the following inclusion criteria:

  * Healthy volunteers aged 18-65 years.
  * The presence of a written and dated informed consent of the volunteer to participate in the program.
  * Consent to observe precautionary measures to limit the circulation of the vaccine virus among people around the vaccinated person (personal hygiene, isolation from unvaccinated children and people with immunodeficiency).
  * Volunteers who are able to fulfill the requirements of the protocol (i.e., fill out a self-observation diary, remember the dates of control visit).

Non-inclusion criteria:

* COVID-19 infection (including cases of asymptomatic carrier).
* Positive test for COVID-19 (PCR).
* Vaccination with any live and / or replicative vaccine one month before screening.
* Neurological disorders that accompany previous vaccination with oral polio vaccine.
* Immunodeficiency condition (primary).
* Malignant neoplasms.
* Immunosuppression (vaccinations are carried out no earlier than 3 months after the end of the course of therapy).
* Pregnancy.
* Hypersensitivity to any component of the vaccine.
* Strong reaction (temperature above 40°C) or a complication on the previous administration of the drug.
* Acute infectious or non-infectious diseases. Vaccinations are carried out 2-4 weeks after recovery or remission. In case of mild acute respiratory viral infections, acute intestinal diseases, vaccinations are carried out after the temperature normalizes.
* The presence in the family or immediate environment (and provided that it is impossible to separate) of unvaccinated against polio (for example, newborns or children who have contraindications to polio vaccinations).
* The presence of persons with immunodeficiency in the family or immediate environment (and provided that it is impossible to separate).

Exclusion Criteria:

* A volunteer can be excluded from the study under the following conditions:

  * Refusal of a volunteer to participate in the program.
  * The need for procedures and / or drug treatment that are not permitted by the protocol of this study.
  * The volunteer was included in violation of the inclusion/non-inclusion criteria of the Protocol.
  * The appearance of non-inclusion criteria during the study.
  * Non-compliance with the research procedures by the volunteer.

    • Any condition of the volunteer that requires, in the reasonable opinion of the research doctor, the withdrawal of the volunteer from the study.
  * The volunteer is out of observation. • For administrative reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be invited to participate in the program. The concept of "healthy" is defined as the absence of deviations detected during the collection of a medical history, during standard clinical and instrumental examinations, as well as in the absence of clinically significant deviations (from the reference values of the laboratory) in laboratory blood and urine tests.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
The number of detected cases | within 12 months by groups
  The number of detected cases confirmed by laboratory (PCR and / or serological tests).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Educational Institution of Higher Education Kirov State Medical University of the Ministry of Health of Russia, Kirov, Russia

REFERENCES:
- [Derived] Yagovkina NV, Zheleznov LM, Subbotina KA, Tsaan AA, Kozlovskaya LI, Gordeychuk IV, Korduban AK, Ivin YY, Kovpak AA, Piniaeva AN, Shishova AA, Shustova EY, Khapchaev YK, Karganova GG, Siniugina AA, Pomaskina TV, Erovichenkov AA, Chumakov K, Ishmukhametov AA. Vaccination With Oral Polio Vaccine Reduces COVID-19 Incidence. Front Immunol. 2022 May 30;13:907341. doi: 10.3389/fimmu.2022.907341. eCollection 2022. PMID 35711442